CLINICAL TRIAL: NCT07068607
Title: Efficacy Comparison of Vonoprazan Combined With Different Antibiotics in Dual Therapy for Helicobacter Pylori Eradication: A Prospective, Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongquan Shi (Other)
Responsible Party: Sponsor-Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20252096-F-1
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Gastritis, Indigestion, Helicobacter Pylori Infection, Gastric Cancer, Peptic Ulcer
MeSH Terms: conditions — Gastritis; Dyspepsia; Stomach Neoplasms; Peptic Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Tetracycline; Minocycline; Bismuth; Clarithromycin; Amoxicillin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vonoprazan - amoxicillin dual therapy (Experimental): Vonorazon 20 mg daily for 14 days # amoxicillin 1000 mg by mouth three time daily for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- Vonoprazan-tetracycline dual therapy (Experimental): Vonorazon 20 mg daily for 14 days # tetracycline 500 mg by mouth three time daily for 14 days
  Interventions: Drug: Vonoprazan; Drug: Tetracycline 500mg tid
- Vonoprazan-minocycline dual therapy (Experimental): Vonorazon 20 mg daily for 14 days # minocycline 100 mg by mouth two time daily for 14 days
  Interventions: Drug: Vonoprazan; Drug: Minocycline
- Bismuth-containing quadruple therapy (Active Comparator): Amoxicillin 1000 mg, clarithromycin 500 mg, vonoprazan 20 mg, and colloidal bismuth tartrate 220 mg, all twice a day for 14 days
  Interventions: Drug: Vonoprazan; Drug: Bismuth; Drug: Clarithromycin 500 mg; Drug: Amoxicillin

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan - amoxicillin dual therapy: Vonorazon 20 mg daily for 14 days # amoxicillin 1000 mg by mouth three time daily for 14 days; Vonoprazan-tetracycline dual therapy:Vonorazon 20 mg daily for 14 days # tetracycline 500 mg by mouth three time daily for 14 days; Vonoprazan-minocycline dual therapy:Vonorazon 20 mg daily for 14 days # minocycline 100 mg by mouth two time daily for 14 days; Bismuth-containing quadruple therapy:Amoxicillin 1000 mg, clarithromycin 500 mg, vonoprazan 20 mg, and colloidal bismuth tartrate 220 mg, all twice a day for 14 days
  Other Names: Vonoprazan - amoxicillin dual therapy
Drug: Tetracycline 500mg tid — Vonoprazan-tetracycline dual therapy:Vonorazon 20 mg daily for 14 days # tetracycline 500 mg by mouth three time daily for 14 days
  Arms: Vonoprazan-tetracycline dual therapy
Drug: Minocycline — Vonoprazan-minocycline dual therapy Vonorazon 20 mg daily for 14 days # minocycline 100 mg by mouth two time daily for 14 days
  Arms: Vonoprazan-minocycline dual therapy
Drug: Bismuth — Bismuth-containing quadruple therapy:Amoxicillin 1000 mg, clarithromycin 500 mg, vonoprazan 20 mg, and colloidal bismuth tartrate 220 mg, all twice a day for 14 days
  Arms: Bismuth-containing quadruple therapy
Drug: Clarithromycin 500 mg — Bismuth-containing quadruple therapy:Amoxicillin 1000 mg, clarithromycin 500 mg, vonoprazan 20 mg, and colloidal bismuth tartrate 220 mg, all twice a day for 14 days
  Arms: Bismuth-containing quadruple therapy
Drug: Amoxicillin — Vonoprazan - amoxicillin dual therapy:Vonorazon 20 mg daily for 14 days # amoxicillin 1000 mg by mouth three time daily for 14 days; Bismuth-containing quadruple therapy:Amoxicillin 1000 mg, clarithromycin 500 mg, vonoprazan 20 mg, and colloidal bismuth tartrate 220 mg, all twice a day for 14 days
  Arms: Bismuth-containing quadruple therapy; Vonoprazan - amoxicillin dual therapy

SUMMARY:
This study aims to evaluate the efficacy of vonoprazan combined with different antibiotics in dual therapy for Helicobacter pylori eradication treatment. Newly infected patients were randomly assigned to four groups: amoxicillin dual therapy, tetracycline dual therapy, minocycline dual therapy, and bismuth quadruple therapy. At the follow - up visit in the 6th week, urea breath test, rapid urease test, or Helicobacter pylori fecal antigen test will be conducted to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 14 days and subjects eligibility will be evaluated after signing informed consent. One of urea breath test#rapid urease test or helicobacter pylori stool antigen test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 14 and 16.

Follow-up: includes one visits. Approximately 28 days after the end of treatment. Eradication of H. Pylori will be confirmed by one of urea breath test#rapid urease test or helicobacter pylori stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 70 years, regardless of gender;
2. Patients with definite Hp infection (positive result in any one of the 13C/14C urea breath test, rapid urease test, and fecal Hp antigen test) who have never received Helicobacter pylori eradication treatment;
3. For women of child - bearing age, it is required to use medically acceptable contraceptive methods during the trial period and within 30 days after the end of the trial.

Exclusion Criteria:

1. Patients who have been definitely diagnosed with Hp infection and have received antibiotic eradication treatment;
2. Patients with contraindications to the study drug or who are allergic to the study drug;
3. Patients with severe organ damage and complications (such as liver cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases;
4. Patients who have been continuously using anti - ulcer drugs (including taking PPI within 2 weeks before the Hp infection test), antibiotics or bismuth complexes (more than 3 times a week within 1 month before screening);
5. Pregnant and lactating women;
6. Patients who have undergone upper gastrointestinal surgery;
7. Patients with moderate or severe atypical hyperplasia or high - grade intraepithelial neoplasia;
8. Patients with symptoms of dysphagia;
9. Patients with evidence of bleeding or iron - deficiency anemia;
10. Patients with a history of malignant tumors;
11. Patients with a history of drug or alcohol abuse within the past 1 year;
12. Patients who are using systemic glucocorticoids, non - steroidal anti - inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except for using aspirin ≤ 100 mg/d);
13. Patients with mental disorders;
14. Patients who have participated in other clinical trials within the past 3 months;
15. Patients who refuse to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication#established by negative [13C] urea breath test #DOB value below 3.9#28 days after the end of eradication

SECONDARY OUTCOMES:
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache,dizziness,skin rash,other gastrointestinal disorders,pyrexia,cough and back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No